CLINICAL TRIAL: NCT01391702
Title: How Sweet is it? Measurement of Glucose in Epidural Fluid and Fluid Obtained During Spinal Anesthesia After a Failed Epidural Using a Bedside Monitor
Brief Title: How Sweet is it? Measurement of Glucose in Epidural and Spinal Fluid
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H11-00901
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Epidural and Spinal Anesthesia for Cesarean Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Labouring woman with epidural in situ: Any healthy English-speaking pregnant woman in labour who has received an epidural for pain relief

SUMMARY:
When a woman requires a cesarean section after labour, anesthesia is usually provided by a pre-existing epidural. Occasionally, the epidural does not work. The anesthesiologist then may give a "spinal anesthetic". The spinal space is identified by seeing cerebrospinal fluid (CSF) in the spinal needle. Rarely a spinal fails after a failed epidural as the fluid seen is epidural space fluid, not CSF. This study plans to use a bedside glucose monitor to measure glucose (sugar) in epidural fluid (compared to CSF) allowing the anesthesiologist to know the spinal needle is in the correct space.

The investigators hypothesize that a bedside glucose measurement device can accurately quantitate the level of glucose within epidural space aspirate, and therefore could aid differentiation between CSF and epidural fluid.

DETAILED DESCRIPTION:
It would be clinically useful to have a bedside test to confirm that the fluid obtained during insertion of a spinal needle following a failed epidural is, in fact, CSF prior to the injection of local anesthetic. This test also may decrease the probability of a failed spinal following a failed epidural top up, and therefore avoid the risks of general anesthesia in the parturient.

When a cesarean delivery is required following a trial of labour, an epidural catheter in situ can be used to provide surgical anesthesia. A large volume (10-20 milliliters) of local anesthetic is administered through the epidural catheter. This is aimed to produce a dense nerve block up to T4 (nipple level), which is sufficient for lower abdominal surgery.

Occasionally, however, this technique does not provide adequate anesthesia for a surgical intervention - termed a 'failed epidural top-up' - and this is estimated to occur up to 38% of the time. Options following the failure of an epidural top-up are dependent on the urgency of delivery, and include either a general anesthetic or an intrathecal injection of local anesthetic (a 'spinal'). The preferred choice for both mother and baby, if time allows, is normally considered to be a spinal.

A spinal is performed by inserting a needle into the subarachnoid space which is surrounded by the epidural space. The subarachnoid space contains CSF, the spinal cord and exiting nerves from the spinal cord. The anesthesiologist identifies the subarachnoid space by obtaining CSF through the needle. Local anesthetic can then be injected directly into the space.

Rarely, spinal anesthesia may fail when administered following a failed epidural, and there are several theories as to why this may occur.

One possible reason for spinal failure is that the large volume of local anesthetic, which is injected down the epidural catheter for cesarean delivery anesthesia, can cause the subarachnoid space to collapse, making it difficult to access with a needle and obtain CSF.

Another theory for failed spinal anesthesia involves misidentification of the clear fluid that returns through the spinal needle. It is postulated that in these circumstances the fluid seen is not CSF. It may be tissue fluid from the epidural space (transudate), local anesthetic that was injected into the epidural space or a combination of the two. In these cases, the needle is not in the subarachnoid space and, therefore, spinal anesthesia will fail.

Anatomical variations, such as a congenital arachnoid cyst, may also contribute to failed spinals following failed epidural top ups.

Various bedside tests have been described to confirm whether the fluid exiting the needle is CSF, including analyzing the fluid's temperature, density, pH, glucose content and whether it precipitated with thiopental (an alkaline solution). Whilst no single test has been completely effective, measurement of glucose seems to be the best indicator. Glucose is thought to be a good discriminator of the fluid obtained through a spinal because of the different proportions of glucose in the clear fluids which could return through the spinal needle. The level of glucose in the CSF is usually approximately 2/3 of plasma glucose (approximately 2-4mmol/L). There should be minimal glucose in the fluid drawn from the epidural space. However, a previous study has shown that a small amount of glucose may be present in the epidural space from 30 minutes after epidural catheter insertion. Potential sources of glucose in the epidural space may be blood, CSF or transudate.

In the past, the presence of glucose was done using a simple reagent strip, which is rapid (2 minutes) and accurate (when compared to laboratory values and testing), however, it solely detects either the presence or absence of glucose. As there may be a small amount of glucose present in the epidural space, the use of reagent strips may not distinguish between epidural fluid and CSF.

A glucose meter gives an absolute value for glucose, which may be more useful. Even though the epidural fluid may contain glucose, the absolute value would be significantly lower than that seen for CSF glucose. The range for normal CSF glucose in the parturient was confirmed using the bedside glucose meters in the Sweet CSF Study as 2-4 mmol/L. In this previous study we compared the efficacy, accuracy and ease of use of three glucose meters that were used to measure CSF glucose.1 The CSF glucose levels were compared to the results from the laboratory measurement of glucose. This study took place January - November, 2010 at BC Women's Hospital in Vancouver, British Columbia. The study established the feasibility of measuring CSF glucose measured with the three glucose meters, and for two meters, verified commonly accepted normal ranges in parturients having elective cesarean delivery under spinal anesthesia.

Now that we have obtained these values, we aim to see if the glucose levels of epidural space fluid (via an epidural catheter) differ from those of CSF using one of the previously tested bedside monitors. We also aim to distinguish the level of glucose in the fluid that returns through the needle if a spinal is done following a failed epidural.

Labouring women admitted to BC Women's will be assessed for eligibility for the study. Women who receive an epidural for labour analgesia will be approached by an investigator who will explain the project and answer questions about the study. Written information regarding the aims and practicalities of the study will be given to women. Informed consent will be obtained following the decision to proceed to cesarean delivery. Women will only be approached for consent to participate if there is time before their surgery. The study will not delay the surgery or interfere with routine standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (American Society of Anesthesiologists (ASA) 1 or 2 classification) with a pre-existing epidural. This will include women with uncomplicated disorders of glucose metabolism e.g. gestational diabetes, insulin dependent gestational diabetes and insulin dependent diabetes.
* Singleton pregnancy
* Age 19 years or older
* Understand written and oral English

Exclusion Criteria:

• Emergency cesarean delivery where time would not allow full consent or sampling

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy pregnant women who are admitted to the hospital in labour who receive an epidural for pain relief
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To confirm that the glucose meter is a feasible and accurate bedside method to detect glucose in epidural aspirate and to use glucose to differentiate CSF from epidural aspirate in women with pre-existing epidural catheters. | Between 2-24 hours after labouring woman has an epidural placed for her labour
  Descriptive statistics outlining the range, central tendency (mean, median), and variability (standard deviation) for epidural glucose will be presented, and these figures then compared to those obtained from the Sweet CSF study.

SECONDARY OUTCOMES:
Influence of other factors on epidural glucose | Between 2-24 hours after labouring woman has an epidural placed for her labour
  Paired t-tests will be conducted to compare epidural glucose levels, blood glucose levels and the influence of the following on the glucose concentration within the epidural aspirate:
  1. Glucose ingestion
  2. Intravenous administration of glucose containing fluids
  3. Disorders of glucose metabolism
  4. Length of time that the epidural catheter was in situ

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Villar, MD, FRCPA, Principal Investigator — University of British Columbia, BC Women's Hospital
Locations (2):
- Canada (2):
  - BC Women's Hospital, Vancouver, British Columbia
  - British Columbia's Women's Hospital, Vancouver, British Columbia